CLINICAL TRIAL: NCT06105125
Title: Periodontal Regeneration in Non-contained Intrabony Defects Using Autologous Micrografts From the Palatal Mucosa: a Randomized Controlled Clinical Trial
Brief Title: Autologous Micrografts From the Palatal Mucosa for Periodontal Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rigenera_Turin
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous micrograft from the palate (Experimental): Modified papilla preservation technique with a combined approach using a bone substitute soaked with autologous micrografts from the palate.
  Interventions: Device: Rigenera + bone substitute
- Control group (Active Comparator): Modified papilla preservation technique with a combined approach using a bone substitute.
  Interventions: Device: Bone substitute alone

INTERVENTIONS:
Device: Rigenera + bone substitute — Minimally invasive flap elevation and debridement of the intrabony defect with micro-curettes. A small punch of connective tissue will be harvested from the palate in the premolar region. Then the graft will be mechanically dissociated using the Rigenera Machine System rotating speed to 80 rpm, in 1.0 ml sterile physiologic solution. After dissociation, the cellular suspension will be passed through a disposable grid with 100 hexagonal blades filtering cells and components of extracellular matrix with a cut-off of 50 um in an average time of 90 s. Finally, part of the suspension containing AMGs will be seeded on the scaffold material and subsequently compacted within the defect. Flaps will be positioned at the pre-surgical level or slightly coronal without any tension.
  Arms: Autologous micrograft from the palate
Device: Bone substitute alone — Minimally invasive flap elevation and debridement of the intrabony defect with micro-curettes. The defect will be filled with the same bone substitute employed in the test group. Finally, flaps will be positioned at the pre-surgical level or slightly coronal without any tension.
  Arms: Control group

SUMMARY:
Some research studies have demonstrated that autologous micrografts made out of different oral tissues may enhance tissue regeneration. The primary aim of this study is to evaluate the clinical performance of a combined approach using an autologous micrograft derived from the palatal mucosa with an alloplastic scaffold for periodontal regeneration of intrabony defects in terms of clinical attachment level gain (primary outcome) and other secondary outcomes (probing pocket depth reduction, radiographic bone fill) compared to a scaffold alone. Moreover, this study aims to compare early wound healing and patient-reported outcome measures between the two groups.

ELIGIBILITY:
Patients selected for the study should fulfil the following inclusion criteria:

* Affected from stage III-IV periodontitis.
* Completed non-surgical periodontal therapy.
* FMPS <15% at 3-month re-evaluation.
* FMBS <15% at 3-month re-evaluation.
* At least one site with an interproximal intrabony defects and residual PPD ≥ 6 mm at re-evaluation, with a radiographic intrabony component ≥ 3 mm, extending to the lingual/palatal side as assessed by preoperative bone sounding.
* Intrasurgically, the defect has to present a non-supporting anatomy (1-2 residual walls in its most coronal portion), requiring flap elevation on both buccal and oral side for its accessibility.
* Signed informed consent.

Exclusion criteria:

* Compromised general health which contraindicates the study procedures (ASA III-VI patients).
* Systemic diseases/medications which could influence the outcome of the therapy (e.g. uncontrolled diabetes mellitus, non-plaque-induced gingival diseases, antiepileptic drugs (phenytoin and sodium valproate), certain calcium channel-blocking drugs (e.g., nifedipine, verapamil, diltiazem, amlodipine, felodipine), immunoregulatory drugs (e.g., cyclosporine), and high-dose oral contraceptives.
* Current smokers (self-reported), users of chewing tobacco, and drug/alcohol abusers.
* Pregnant or nursing women.
* Presence of furcation involvement ≥ II degree (Hamp 1975) at the affected teeth.
* Very large and wide defects that required the use of membrane.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level change | 12 months
  Clinical attachment level will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Probing pocket depth change | 12 months
  Probing depth will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Radiographic bone level change | 12 months
  Periapical standardized radiographs will be taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)
Patient reported outcome measures | 2 weeks
  Pain will be self-recorded by the patient using a visual analog scale (from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy